CLINICAL TRIAL: NCT07176429
Title: Pseudoaccommodation of the Light Adjustable Lens: A Comparative Study
Brief Title: Pseudoaccommodation of the Light Adjustable Lens: A Comparitive Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Helm Vision Group (Other)
Responsible Party: Principal Investigator, Craig J. Helm, President, Helm Vision Group, Helm Vision Group
Other Study IDs: 2025-0503
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Amplitude of Pseudoaccommodation
Keywords: Pseudoaccommodation, light adjustable lens, monofocal lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Participants who have had the Light Adjustable Lens implanted with cataract surgery: Participants who have had the Light Adjustable Lens Plus implanted surgically
  Interventions: Device: Measurement of refractive error and amplitude of pseudoaccommodation
- Participants who have had the Akreos AO60 lens implanted with cataract surgery
  Interventions: Device: Measurement of refractive error and amplitude of pseudoaccommodation
- Participants who have had the Light Adjustable Lens Plus implanted
  Interventions: Device: Measurement of refractive error and amplitude of pseudoaccommodation

INTERVENTIONS:
Device: Measurement of refractive error and amplitude of pseudoaccommodation — We will be using an assessor, masked as to which participant received what particular lens implant to determine the range of pseudoaccommodation in each eye. This will be done for each eligible eye and the 3 cohorts will be studied and compared.
  Other Names: Measurement of pupillary size; Measurement of spherical aberration of the eye

SUMMARY:
Cataract surgery involves the removal of a cloudy natural lens, followed by the implantation of an artificial lens. The choice of lens implant helps determine what the vision will be like after surgery. "Monofocal" lens implants are not designed to give both distance and close-up vision at the same time. We wish to study the amount of reading ability that a lens implant corrected for distance vision will provide. Eligible study participants include those who have had cataract surgery with implantation of either the Light Adjustable Lens® (LAL), the Light Adjustable Lens Plus® (LAL+) or the Bausch & Lomb Akreos® AO60 lens implant. We anticipate enrolling up to 100 subjects in this study.

These lens implants are designed to achieve excellent distance vision, inasmuch as the lens implant target is achieved. The lens implant target of excellent, unaided distance vision is more likely to be achieved when the chosen power of the lens implant matches the eye's curvature and length. Before cataract surgery, the eye is measured by a machine, and the information is used to calculate which lens power is predicted to best match the eye. In the case of the LAL, a light delivery device is used after surgery to fine-tune the power of the lens implant and achieve sharper unaided vision.

Although both of these lens implants are technically "monofocal" lenses and work well for distance vision, they differ in ways that affect near vision. "Pseudoaccommodation" is the term that refers to the ability of an eye with a lens implant to see up close without glasses. The optical qualities of the Light Adjustable Lens generally allow eyes implanted with this lens to see objects at an intermediate or close-up range without glasses. The amount of pseudoaccommodation or close-up ability in these eyes differs from person to person.

The purpose of this study is to determine the average amount of reading ability in eyes implanted with the Light Adjustable Lens® and compare it to the amount measured with the Bausch & Lomb AO60 lens.

DETAILED DESCRIPTION:
The purpose of this study is to measure the capability of three different monofocal (non-multifocal) lens implants to also provide near vision when corrected for distance vision. We will be comparing two versions of the Light Adjustable Lens® (RxSight, Irvine, CA) and also the Akreos® AO60 lens (Bausch & Lomb, Bridgewater, NJ). All three of these lens FDA-approved lens implants were categorized as being "monofocal", meaning that all light rays entering the eye are focused at one particular point. This means that when eyes that have these types of lens implants are corrected to see well at distance, that the near vision should be poor (when not wearing bifocals or other glasses to specifically aid near vision. The Light Adjustable Lenses are touted as having an unusually high ability to deliver reading vision in addition to distance vision, despite being a monofocal lens. We aim to determine what the range of near vision is (defined as "pseudoaccommodation") for the Light Adjustable Lens, the Light Adjustable Lens Plus, and the Akreos® AO60 lens. We have not found this information available on a PubMed search. This information would be very useful clinically for counselling patients prior to cataract surgery. It would also help determine if there is a correlation between those who end up having a high degree of pseudoaccommodation and other factors such as pupil size and total amount of spherical aberration of the eye (which is thought to influence near vision).

Cataract surgery consists of the removal of the natural crystalline lens of the eye when the lens becomes cloudy. To restore the focusing power of the eye, an artificial lens is typically implanted immediately after cataract removal, during the same operation. The lens implants are made in a range of powers that allow selection of a power that corrects the refractive error of the eye and reduces or eliminates the need for glasses or contact lenses. The Light Adjustable Lens® (LAL) by RxSight is the world's only lens implant that allows the lens implant power to be adjusted or fine-tuned after it's been implanted into the eye.

"Accommodation" is the process by which the natural lens is changed in shape and position to allow a person to see both far and near without glasses. This ability is gradually lost, usually beginning in the mid-40s, when a person starts to develop a need for reading glasses. This happens as the natural crystalline lens begins to lose its elasticity. The Helmholtz theory is the most widely held theory for how accommodation works. It holds that the effort to see near objects causes contraction of the ciliary body in the eye. The crystalline lens is attached to the ciliary body via zonules or fibers. Thus, when the ciliary body contracts, the tension on the zonules loosens, allowing the lens to thicken and shift forward in position. These changes increase the focusing power of the eye. Therefore, when the lens loses its elasticity, it becomes less able to thicken and increase its focusing power. When cataract surgery is performed and a lens implant is placed, because the lens implant is rigid, true accommodation is lost. However, some ability to see both distant objects and near objects is maintained to some degree. This ability to see both far and near in an eye that has had a lens implant placed is called "pseudoaccommodation". Pseudoaccommodation can result from a combination of factors, including forward movement of the lens implant with contraction of the ciliary body, pupil size, and residual spherical aberration of the eye. "Spherical aberration" is a type of optical distortion that occurs because with a curved surface, light rays are focused either more strongly (positive spherical aberration) or less strongly (negative spherical aberration) as the rays pass through the surface further away from its center. This means that not all light rays are focused at one point. Rather, a range of reduced sharpness is produced, resulting in a range of less clear vision, instead of a single focal point of clarity.

In addition to its ability to be adjusted to fine-tune distance vision, the LAL is associated with increased near vision in subjects who also have good distance vision. In other words, this lens implant seems to provide a higher-than-normal degree of pseudoaccommodation compared to other monofocal (non-multifocal) lens implants. Although encountered in clinical practice, the reasons for this high degree of pseudoaccommodation are complicated. It is believed, in part, to be related to the shape of the lens implant, which produces negative spherical aberration. Clinically, the reading ability of recipients of the lens varies from person to person. This may be partly related to the differing amounts of residual spherical aberration that are left in the eye after the LAL has been adjusted with the light delivery device to fine-tune the visual acuity.

ELIGIBILITY:
Inclusion Criteria: Those who have had cataract surgery with implantation of either the Light Adjustable Lens or the Light Adjustable Lens Plus, or the Akreos AO60 lens implants. Must have not had previous keratorefractive surgery and no ocular pathology that precludes being correctable to 20/20 vision.

-

Exclusion Criteria: Those under 18 years of age, those unable to give informed consent, prisoners, or those who are pregnant.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those who have had cataract surgery with the Light Adjustable Lens, the Light Adjustable Lens Plus, or the Akreos AO60 lens implant.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Amplitude of pseudoaccommodation | 1 day
  Range of near-vision as measured through best distance correction

CONTACTS AND LOCATIONS:
Locations (1):
- Helm Vision Group, Valencia, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We can share our raw data from our spreadsheet.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2026 through May 2031
Access Criteria: The PI and study coordinator will have access to the collated data on the spreadsheet.